CLINICAL TRIAL: NCT00775242
Title: Comparative Efficacy and Safety Study of Three Different Doses of a Formulation Composed of Crystalline Estradiol and Progesterone Microspheres, Indicated for Monthly IM Injection for the Treatment ot Climacteric Symptoms.
Brief Title: Efficacy and Safety of Estradiol and Progesterone Microspheres for the Treatment of Climacteric Symptoms.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centro A.F. de Estudios Tecnologicos, S.A. (Industry)
Responsible Party: Juan Angeles Uribe, Centro A.F. de Estudios Tecnológicos, S.A.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02/PAF/06; 0607/I/APL
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Menopause
Keywords: Menopause; Hormone Replacement Therapy; Microspheres; Progesterone; Estradiol; Hot flashes
MeSH Terms: conditions — Hot Flashes | interventions — Estradiol; Progesterone; Estrogens; Progestins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Estradiol and progesterone injection (Experimental): Comparison of three different dosages of estradiol and progesterone a) 0.5 mg E/15 mg P; b) 1 mg E/20 mg P; c) 1 mg E/30 mg P
  Interventions: Drug: Estradiol and Progesterone

INTERVENTIONS:
Drug: Estradiol and Progesterone — Injectable suspension of three different dosages of estradiol and progesterone a) 0.5 mg E/15 mg P; b) 1 mg E/20 mg P; c) 1 mg E/30 mg P. Administered on a monthly basis during a six-month period.
  Other Names: estrogens and progestines
Drug: Estradiol and Progesterone — Injectable suspension of three different formulations of estradiol and progesterone a) 0.5 mg E/15 mg P; b) 1 mg E/20 mg P; c) 1 mg E/30 mg P. Each will be applied on a monthly basis during a six-month period
  Other Names: Estrogens; Progestins

SUMMARY:
During menopause a woman's body slowly produces less of the hormones estrogen and progesterone. Lower hormone levels in menopause may lead to hot flashes, vaginal dryness and osteoporosis. To help with these problems, women are often given estrogen or estrogen with progestin. The purpose of this study is to assess and compare the efficacy and safety of three doses of estradiol and progesterone for the treatment of the climacteric symptoms

DETAILED DESCRIPTION:
Different formulations of estrogens and progestins have been used for the treatment of climacteric symptoms, however up to this date no formulation is completely satisfactory. Our company has developed a new technology for the preparation of controlled release bioerodible non-polymeric microspheres, these microspheres are capable of delivering doses of estradiol (E) and progesterone (P) at levels appropriate for the Hormonal Replacement Therapy (HRT) in order to relieve the climacteric symptoms. Non clinical and clinical studies have been conducted aimed at assessing the pharmacokinetics of these microspheres, at several doses of progesterone and estradiol. Results show that sustained plasma profiles for both steroids within the therapeutic range for several days are attained. On this basis, a new efficacy and safety study is going to be conducted with the purpose of assessing and defining the most appropriate doses of estradiol and progesterone for the HRT of the climacteric symptoms.

Three different doses of progesterone and estradiol (0.5 mg of E + 15 mg of P vs 1 mg of E + 20 mg of P vs 1 mg of E + 30 mg of P) will be compared in terms of their efficacy and safety to treat the climacteric symptoms in healthy postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 65 years.
* Perimenopausal subjects: Women showing spontaneous amenorrhea during the last 11 months.
* Postmenopausal subjects: Women with not less than 12 consecutive months of amenorrhea and FSH > 40 mIU/mL
* Subjects showing vasomotor symptoms, not less than 3 hot flashes in a day or not less than 21 hot flashes in a week
* Healthy subjects determined on the basis of a satisfactory complete clinical history, clinical laboratory tests, cervical cytology, endometrium biopsy and vaginal pelvic ultrasonography.
* Subjects not receiving any hormonal treatment.

Exclusion Criteria:

* Subjects with background of endometrial hyperplasia or endometrial cancer.
* Subjects with endometrial hyperplasia or endometrial cancer assessed by endometrial biopsy.
* Perimenopausal subjects with background of abnormal uterine bleeding unless the Principal Clinical Investigator considers that this abnormality is secondary to the menopausal condition.
* Subjects with hypersensitivity to any medicament.
* Subjects with direct family background of breast cancer.
* Subjects with background of cardiovascular disease, renal, hepatic, metabolic, gastrointestinal, neurologic, endocrine, gynecologic disease including dysfunctional uterine bleeding, cervico uterine dysplasia, cancer, anemia, emotional disorders, or any other chronic degenerative disorders which could affect her participation in the study.
* Subjects who require any medicament in the course of the study unless the Principal Clinical Investigator considers that there is no pharmacological interaction.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2007-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change of frequency and intensity of vasomotor symptoms | 0, 1, 2, 3, 4, 5, 6 and 7 months

SECONDARY OUTCOMES:
Frequency and intensity of vulvar and vaginal atrophy symptoms Vaginal pH Index of vaginal maturation (surface, intermediate and parabasal cells) Karyopiknotic index Lipids profile Utian quality of life scale Green climacteric symptoms scale | 0, 1, 2, 3, 4, 5, 6 and 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Cortes Bonilla, Ob/Gyn, Principal Investigator
Locations (1):
- Centro A.F. de Estudios Tecnologicos, S.A., Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Cortes-Bonilla M, Alonso-Campero R, Bernardo-Escudero R, Francisco-Doce MT, Chavarin-Gonzalez J, Perez-Cuevas R, Chedraui P. Improvement of quality of life and menopausal symptoms in climacteric women treated with low-dose monthly parenteral formulations of non-polymeric microspheres of 17beta-estradiol/progesterone. Gynecol Endocrinol. 2016 Oct;32(10):831-834. doi: 10.1080/09513590.2016.1183628. Epub 2016 May 17. PMID 27187320